CLINICAL TRIAL: NCT01587664
Title: Safety and Efficacy Evaluation of the NewBreez Intra-laryngeal Prosthesis
Brief Title: NewBreez Safety and Efficacy Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of recruitment and loss of the French principal investigator.
Sponsor: ProTiP Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIL-02-PEC-1-A
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Swallowing Disorders
Keywords: Swallowing disorders; Aspiration
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NewBreez ILP (Experimental): Implantation of a NewBreez ILP
  Interventions: Device: NewBreez ILP

INTERVENTIONS:
Device: NewBreez ILP — NewBreez ILP implantation

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of the NewBreez intra-laryngeal implant in patients with dysfunctional larynx.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Congenital or acquired, central or peripheral, neurological or neuromuscular disorder associated with laryngeal dysfunction with aspirations
3. Has a tracheotomy or tracheostomy and is indicated for use of a hood weaning kit
4. Must be able to comply with all study requirements for the duration of the study as outlined in the protocol. This includes complying with the visit schedule as well as study specific procedures such as: scanner, radiographic swallowing study, nasopharyngoscopy , NewBreez ILP implant as well as quality-of-life evaluation
5. Must be able to understand and be willing to provide written informed consent

Exclusion Criteria:

1. Any condition that precludes the insertion of the NewBreez ILP or ancillary implantation device
2. Major swallowing disorder
3. Existing coagulation disorder
4. Previous esophageal stenting
5. Life-expectancy < 12 months
6. Be pregnant or breastfeeding or intention of becoming pregnant during the study (if female of childbearing potential)Point of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Aspiration score at 1 month | 1 month
  Within-subject relative change-from-baseline at 1 month in aspiration score based on radiographic swallowing study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Remacle, Prof., Principal Investigator — UCL Mont-Godinne (Belgium)
Locations (2):
- CHU Mont-Godinne, Yvoir, Belgium
- Hopital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No